CLINICAL TRIAL: NCT03707691
Title: Pitch Perception and Memory: Deficits and Training
Acronym: Pitch_Train
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0632; 2018-A02670-55 (Other: ID-RCB)
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-04

CONDITIONS: Cochlear Implants
Keywords: Hearing; Cochlear Implants; Congenital Amusia; Pitch; Audio-visual interactions
MeSH Terms: conditions — Tune Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cochlear implant users (Experimental): In both arms a pitch training protocol and a visuo-spatial training protocol are applied.
  Interventions: Behavioral: Listening tests. Pitch training protocol; Behavioral: visuo-spatial training protocol; Behavioral: EEG/MEG/MRI recordings.
- Participants with Congenital Amusia (Experimental): In both arms a pitch training protocol and a visuo-spatial training protocol are applied.
  Interventions: Behavioral: Listening tests. Pitch training protocol; Behavioral: visuo-spatial training protocol; Behavioral: EEG/MEG/MRI recordings.
- Control Participants (Experimental)
  Interventions: Behavioral: Listening tests. Pitch training protocol; Behavioral: visuo-spatial training protocol; Behavioral: EEG/MEG/MRI recordings.

INTERVENTIONS:
Behavioral: Listening tests. Pitch training protocol — The two training protocols consists of perceptual tasks (auditory or visual exercises) performed repetitively using a tablet. Each protocol consists in 30 sessions of ~20 minutes performed at home over a period of 15 weeks.
Behavioral: visuo-spatial training protocol — The two training protocols consists of perceptual tasks (auditory or visual exercises) performed repetitively using a tablet. Each protocol consists in 30 sessions of ~20 minutes performed at home over a period of 15 weeks.
Behavioral: EEG/MEG/MRI recordings. — Listening tests. EEG/MEG/MRI recordings

SUMMARY:
Pitch perception and memory are central in auditory cognition, in particular for sound source segregation and recognition, speech prosody and music processing. Here the investigator assess pitch perception and memory in hearing-impaired listeners wearing cochlear implant(s) and listeners with congenital amusia, both compared with control listeners. Behavioral, EEG, and MEG measures are collected in audio and audio-visual contexts to characterize pitch processing deficits, and test a pitch training program.

ELIGIBILITY:
Inclusion Criteria:

For adult participants:

* Aged between 18 and 90
* Absence of neurological and psychiatric disorders
* No major cognitive deficit, ability to understand and apply study instructions
* Motivation to participate efficiently in the study
* Written informed consent to participant in the study
* Affiliated to social security
* Control participants and participants with congenital amusia for Experiment 5: MRI/MEG compatibility

For underage participants:

* Subject aged 5 years and over
* Informed consent of parents or guardians for the participation of the child being studied
* No neurological or psychiatric history
* Without major cognitive impairment and ability to understand and apply setpoint.
* Subject affiliated to a social security scheme
* Motivation to participate effectively in the project

Exclusion Criteria:

For adult participants:

* Age below 18 or above 90
* Pregnant or breast-feeding woman

For underage participants:

- Pregnant or nursing minors

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2027-10-26 (Estimated); Study Completion 2027-10-26 (Estimated)

PRIMARY OUTCOMES:
percentages of correct responses in listening tests | during procedure
reaction times in listening tests | during procedure
Event-Related Fields | during procedure
  MEG measurements
Oscillations | during procedure
  MEG measurements

SECONDARY OUTCOMES:
percentages of correct responses | Day 0
  Performance in listening tests in audio contexts
percentages of correct responses | Day 0
  Performance in listening tests in audio-visual contexts
reaction times | Day 0
  Performance in listening tests in audio contexts
reaction times | Day 0
  Performance in listening tests in audio-visual contexts
Event-Related Fields | Day 0
  EEG measurements
Oscillations | Day 0
  EEG measurements

CONTACTS AND LOCATIONS:
Overall Officials: Anne CACLIN, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Lyon Neuroscience Research Center, Bron, France

IPD SHARING:
Plan to Share IPD: No